CLINICAL TRIAL: NCT02050555
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Evaluate the Effect of Koji-extracted Beverage Fermented With Pediococcus Pentosaceus LP28
Brief Title: Anti-obesity Effect of Koji-extracted Beverage Fermented With Pediococcus Pentosaceus LP28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Marukome Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-867
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Koji-extracted beverage (Placebo Comparator): 100ml/day for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Koji-extracted beverage fermented with LP28 (Experimental): 100ml/day for 12 weeks. 1x10^11 cells (LP28)/day
  Interventions: Dietary Supplement: Koji-extracted beverage fermented with Pediococcus pentosaceus LP28

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Koji-extracted beverage
Dietary Supplement: Koji-extracted beverage fermented with Pediococcus pentosaceus LP28
  Arms: Koji-extracted beverage fermented with LP28

SUMMARY:
This study is designed to evaluate the effect of koji-extracted beverage fermented with Pediococcus pentosaceus LP28 on BMI and body fat in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-30 kg/m2

Exclusion Criteria:

* Taking drugs or functional food that may affect body weight or body fat
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease
* History of severe disease and/or major surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in BMI from baseline | Every 4 weeks (Overall 12 weeks)
Change in body fat mass (percentage) from baseline | Every 4 weeks (Overall 12 weeks)

SECONDARY OUTCOMES:
Change in abdominal circumference from baseline | Every 4 weeks (Overall 12 weeks)
Change in visceral fat area by CT scan from baseline | Weeks 0 and 12
Change in 2h glucose concentration after the oral glucose tolerance test (OGTT) from baseline | Weeks 0 and 12
Change in fasting plasma glucose from baseline | Every 4 weeks (Overall 12 weeks)
Change in serum triglyceride from baseline | Every 4 weeks (Overall 12 weeks)
Change in serum total cholesterol from baseline | Every 4 weeks (Overall 12 weeks)
Change in serum LDL cholesterol from baseline | Every 4 weeks (Overall 12 weeks)
Change in serum HDL cholesterol from baseline | Every 4 weeks (Overall 12 weeks)
Change in fasting insulin from baseline | Weeks 0 and 12
Change in homeostasis model assessment-insulin resistance (HOMA-R) from baseline | Weeks 0 and 12
  HOMA-R is calculated as fasting insulin (mU/mL) x fasting glucose (mg/dL) / 405

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan